CLINICAL TRIAL: NCT00124605
Title: Phase I Trial of Arsenic Trioxide in Combination With Pamidronate Disodium
Brief Title: Arsenic Trioxide and Pamidronate in Treating Patients With Advanced Solid Tumors or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03082; PHI-45; U01CA062505 (NIH); CDR0000434807 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Multiple Myeloma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Multiple Myeloma | interventions — Pamidronate; Arsenic Trioxide

ARMS (1):
- Treatment (pamidronate disodium and arsenic trioxide) (Experimental): Patients receive pamidronate IV and over 2 hours on days 1 and 15 and arsenic trioxide IV over 2 hours on days 1-5 and 15-19. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pamidronate disodium; Drug: arsenic trioxide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: pamidronate disodium — Given IV
  Other Names: Aminomux; APD; Aredia; GCP-23339A
Drug: arsenic trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid Anhydride; AS2O3; Trisenox
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy, such as arsenic trioxide and pamidronate, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Arsenic trioxide and pamidronate may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Pamidronate may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving arsenic trioxide together with pamidronate may kill more cancer cells. This phase I trial is studying the side effects and best dose of arsenic trioxide and pamidronate in treating patients with advanced solid tumors or multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the toxicities of the combination of arsenic trioxide in combination with pamidronate disodium at four dose levels.

II. To assess the pharmacokinetics of pamidronate disodium when given in combination with arsenic trioxide.

III. Utilizing 2-color immunofluorescence (IF) to determine if the treatment with combination of arsenic trioxide and pamidronate disodium affects the phosphorylation of epidermal growth factor receptor (EGFR) IV. In patients with multiple myeloma utilizing western blot to evaluate the pre- and post-treatment levels of protein tyrosine phosphatase 1B in lysates of multiple myeloma cells.

V. To obtain preliminary data for response to this regimen in this patient population.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive pamidronate IV and over 2 hours on days 1 and 15 and arsenic trioxide IV over 2 hours on days 1-5 and 15-19. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pamidronate and arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: Approximately 12-24 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven diagnosis of solid tumors or multiple myeloma refractory to standard therapy or for which no satisfactory treatment exists at the time of enrollment
* Patient must be capable of understanding the nature of the trial and must give written informed consent
* Patients must have a WHO performance status of 0, 1, or 2
* Patients must have life expectancy of at least three months
* Absolute neutrophil count of > 1x10^9 /L
* Platelet count > 75 x 10^9 /L
* Calculated creatinine clearance of > 50 mL/min
* Serum bilirubin =< 1.5 x the institutional upper limit of normal
* SGOT (AST) and SGPT (ALT) must be =< 2.5 x the institutional upper limit of normal
* All patients must be willing to use adequate contraception
* Patients with brain metastases which at the time of study enrollment are controlled and do not require treatment with corticosteroids are eligible
* Patients must not have a prolonged QT interval > 460 milliseconds on baseline ECG in the presence of normal serum potassium and magnesium values; ECG must be obtained within 28 days prior to registration
* Patients must not be receiving or planning to receive drugs known to prolong the QT interval
* Patients previously or currently treated with pamidronate or other bisphosphonates are eligible after a wash-out period of 28 days; concurrent treatment with other bisphosphonates is not allowed
* Patients must not have a history of torsades de pointes type ventricular arrhythmia

Exclusion Criteria:

* Patients who have had radiotherapy or chemotherapy within three weeks (nitrosoureas or mitomycin C within six weeks) prior to anticipated first day of dosing; patients must be fully recovered from the acute effects of any prior chemotherapy or radiotherapy
* Patients with uncontrolled electrolyte imbalance (NA < 132 mmol/L; K < 3.5 mmol/L; Mg < 1.7 mg/dL)
* Patients undergoing therapy with other investigational agents; patients must have recovered from all acute effects of previously administered investigational agents and sufficient time must have elapsed since last administration to ensure the drug interactions not occur during this study
* Patients who are pregnant or breast-feeding will be excluded
* Patients with history of hypersensitivity to pamidronate or other bisphosphonates
* Patients previously treated with arsenic trioxide are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest dose tested in which greater than 33% of patients experienced dose limiting toxicity (DLT) assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 28 days
  The toxicities observed at each dose level will be summarized in terms of type, severity, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course. Tabular and graphical summaries will be used to explore the relationship of type and grade of toxicity to dose, course, and pharmacokinetics.

SECONDARY OUTCOMES:
Survival | Up to 4 years
Time to failure | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw Twardowski, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States